CLINICAL TRIAL: NCT03616158
Title: Change in Serum and Sputum Biomarkers Over Time in the Development of Rheumatoid Arthritis-associated Lung Disease
Brief Title: Investigate the Development and Progression of Lung Disease in Rheumatoid Arthritis Over Time
Acronym: RA-LD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: HS-3161
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Rheumatoid Arthritis; Lung Diseases
Keywords: Rheumatoid arthritis; Interstitial Lung Disease; RA; ILD
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and sputum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pre-RA: Subjects with interstitial lung disease (ILD) or airways disease, no rheumatoid arthritis (RA), and positive antibodies will participate in 5 in-person study visits. Additionally, quality of life questionnaires will be mailed/emailed and completed at home every 6 months, at 4 different time points. Overall participation will take place over a 4 year time frame and an additional 6 years of survival follow-up.
  In-person Study Assessments Include:
  1. Medical History and Physical Exams
  2. Quality of Life Questionnaires
  3. Collection of blood
  4. Radiology
  5. Lung Function Test
  6. 6 Minute Walk Test
  7. Bronchoscopy (Clinically indicated)
  8. Sputum (Optional)
  9. Musculoskeletal ultrasound (Optional)
- RA without LD: Subjects with rheumatoid arthritis (RA), and no interstitial lung disease (ILD) or airways disease, will participate in 5 in-person study visits. Additionally, quality of life questionnaires will be mailed/emailed and completed at home every 6 months, at 4 different time points. Overall participation will take place over a 4 year time frame and an additional 6 years of survival follow-up.
  In-person Study Assessments Include:
  1. Medical History and Physical Exams
  2. Quality of Life Questionnaires
  3. Collection of blood
  4. Radiology
  5. Lung Function Test
  6. 6 Minute Walk Test
  7. Bronchoscopy (Clinically indicated)
  8. Sputum (Optional)
  9. Musculoskeletal ultrasound (Optional)
- RA-LD: Subjects with rheumatoid arthritis (RA) and interstitial lung disease (ILD) or airways disease, will participate in 5 in-person study visits. Additionally, quality of life questionnaires will be mailed/emailed and completed at home every 6 months, at 4 different time points. Overall participation will take place over a 4 year time frame and an additional 6 years of survival follow-up.
  In-person Study Assessments Include:
  1. Medical History and Physical Exams
  2. Quality of Life Questionnaires
  3. Collection of blood
  4. Radiology
  5. Lung Function Test
  6. 6 Minute Walk Test
  7. Bronchoscopy (Clinically indicated)
  8. Sputum (Optional)
  9. Musculoskeletal ultrasound (Optional)
- LD Controls: Subjects with interstitial lung disease (ILD) or airways disease, no rheumatoid arthritis (RA), and negative antibodies will participate in 5 in-person study visits. Additionally, quality of life questionnaires will be mailed/emailed and completed at home every 6 months, at 4 different time points. Overall participation will take place over a 4 year time frame and an additional 6 years of survival follow-up.
  In-person Study Assessments Include:
  1. Medical History and Physical Exams
  2. Quality of Life Questionnaires
  3. Collection of blood
  4. Radiology
  5. Lung Function Test
  6. 6 Minute Walk Test
  7. Bronchoscopy (Clinically indicated)
  8. Sputum (Optional)
  9. Musculoskeletal ultrasound (Optional)

SUMMARY:
The purpose of this study is to investigate the link between the lungs and rheumatoid arthritis (RA). Additionally, to understand why RA patients get lung disease, how to treat, and prevent the disease.

DETAILED DESCRIPTION:
This study is to learn more about the risk factors for the development of lung disease among patients with rheumatoid arthritis (RA), an auto-immune disease. Additionally, those at heightened risk of developing RA such as in the pre-RA period. This is a prospective and retrospective study, which 420 patients will be enrolled into the study. In-person participation will be up to 4 years, completing different standard of care assessments yearly. Additionally, quality of life questionnaires will be completed every 6 months at 4 time points. Lastly, an extended follow-up will be performed yearly for an additional 6 years, an overall 10 year participation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80 years

Exclusion Criteria:

1. Subjects who do not speak English
2. Subjects without the capacity to sign the informed consent form (ICF)
3. Pregnant women

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects are selected for participation in the study because they are diagnosed with or without rheumatoid arthritis and lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2023-05-10 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Define which patients with RA (or pre-RA) are at greatest risk for developing RA-related lung disease (LD). | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Solomon, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States